CLINICAL TRIAL: NCT07346560
Title: Primary Versus Secondary Internal Limiting Membrane Peeling in Uncomplicated Retinal Detachment
Brief Title: 1ry Versus 2ry ILM Peeling in RD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaa Abdalsadek Ahmed Sinjab, Lecturer of Ophthalmology, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Soh-Med-25-12-8PD
Record Dates: First submitted 2026-01-06; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Retinal Detachment Rhegmatogenous; ILM Peeling
Keywords: Retinal detachment; ILM peeling; Proliferative vitroretinopathy
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Primary ILM peeling) (Active Comparator): ILM peeling during PPV for rRD
  Interventions: Procedure: Primary ILM peeling
- Group B (Active Comparator): ILM peeling at time of silicon oil extraction
  Interventions: Procedure: Secondary ILM peeling

INTERVENTIONS:
Procedure: Primary ILM peeling — ILM peeling during the 1st surgical intervention for rRD
  Arms: Group A (Primary ILM peeling)
Procedure: Secondary ILM peeling — ILM peeling is delayed for the time of silicon oil extraction
  Arms: Group B

SUMMARY:
Patients with uncomplicated rhegmatogenous retinal detachment will be recruited. All eyes will underwent 23G PPV with silicon oil tamponade. The eyes will be classified into two groups according to the timing of ILM peeling. Group A, ILM peelin will be performed during the first intervention, while in group B, it will be done at the time of silicon oil extraction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with uncomplicated rhegmatogenous retinal detcahment.

Exclusion Criteria:

* PVR
* Recurrent RD
* Tractional RD
* Macular hole RD
* Scleral buckling is indicated
* Macular scarring
* Previous PPV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of complications | From enrollment till 3 months postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag Faculty of Medicine, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be available for other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From enrollment and forever.